CLINICAL TRIAL: NCT03450174
Title: Effectiveness of Multiple Micro-nutrient Fortified Fudge on Nutritional Status of 3-5 Years of Age Children: A Randomize Control Trial
Brief Title: Effectiveness of Multiple Micro-nutrient Fortified Fudge on Nutritional Status of 3-5 Years of Age Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Collaborators: Sindh Lady Health Worker Program for Family Planning and Primary Health Care (Unknown); PCSIR Laboratories Complex Karachi Pakistan (Unknown)
Responsible Party: Principal Investigator, Fakhar Gulzar, PhD Scholar, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: UniversityVAS
Record Dates: First submitted 2018-01-25; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Micronutrient Deficiencies; Anemia; Fortification; Undernutrition; Early Childhood Development
MeSH Terms: conditions — Anemia; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): this group, only placebo product will be given
  Interventions: Dietary Supplement: Placebo
- Formative messages (Experimental): this group will be received only daily formative messages on diet diversity, healthy and best nutrition practices
  Interventions: Behavioral: Formative messgaes
- Fortified product (Experimental): this group will be received only fortified product on alternate day up to 6 months
  Interventions: Dietary Supplement: Fortified product
- Fortified product plus (Experimental): this group will receive fortified product along with daily messages on diet diversity and healthy nutrition practices
  Interventions: Combination Product: Fortified product plus

INTERVENTIONS:
Dietary Supplement: Placebo — In control group, participants will receive only a placebo product
  Arms: Control
Behavioral: Formative messgaes — In this group, participants will only receive daily formative messages
  Arms: Formative messages
Dietary Supplement: Fortified product — In this group, participants will receive fortified product on alternate day up till 8 months
  Arms: Fortified product
Combination Product: Fortified product plus — In this group participants will receive fortified product on alternate day and formative messages up till 8 months
  Arms: Fortified product plus

SUMMARY:
Multiple micro-nutrient deficiencies in Pakistan is wide spread, there is dire need to address these by using smart solutions, among them multiple fortified product (fudge) is an alternate possible way to address this issue. Fortified products have the potential to reduce micronutrient deficiencies in children, therefore in current study children from 3-5 years will receive fortified product along with enhance nutrition promotional information to bring change in their dietary practices and nutritional indices.

DETAILED DESCRIPTION:
As per the National Nutrition Survey, 2011 anaemia (iron deficiency) affected the children severely as one in three children under the age of 5 anemic, whereas prevalence of vitamin A deficiency among children under 5 years is more than 50%, similarly Zinc deficiency children and vitamin D deficiency prevalence in children is more than 40%.

The numerous indicators of nutrition deficiencies are related to inadequately nutritious and safe food, illiteracy, malpractices along with lack of nutritional knowledge and other social and behavioral issues. A healthy and supportive nutritional status, direct toward better intellect and earning of individual, which boost the social impact and macro level change.

Childhood stunting and deficiencies in iron and iodine hamper cognitive development, school achievement and adult productivity by 2.5-19.8 percent subsequently adult anemia reduces work performance in manual labor in the agriculture area and overall resultant US$ 7.6 billion annually loss for Pakistan, which corresponds to nearly 3 percent of GDP all due to poor nutritional indicators, which are preventable. Therefore, in developing countries like Pakistan, robust need is required, to do evidence base and translational research which could be easily converted into action that improves nutritional status.

Food fortification with micro-nutrients is effective, cost-efficient and medium-term approach to improve micro-nutrient status of vulnerable groups and is sustainable once established to prevent these at cheaper cost. There is need to investigate the positive effects of multiple micronutrient administration on child development along with there is dire need for more research to investigate it comprehensively at community level.

Fortified food products such as (milk, wheat, rice, oil, and other) are already in existing strategies worldwide to prevent micro-nutrient deficiencies in society which is well established and currently there are several extensive activities are implemented to prevent these hidden hunger but required results are not achieved.

On the other hand, other smart solutions are emerging to prevent these deficiencies at wider level in best possible means, among them fortified candy with multiple micronutrients is one vehicle. Confectionery products have the potential to carry the micronutrient for better delivery and doesn't significantly affect the flavour, taste and texture of the product.

The objective of the study is to determine the nutritional status, factor causing micronutrient deficiencies in pre-school children in semi-urban area of Karachi and how fortified product and enhance nutritional knowledge can bring change in nutritional indicators and understanding of nutrition in community.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years of age
* no medical complication
* from middle-income group within the semi-urban population

Exclusion Criteria:

* illness/ infections (TB, Malarial drug)
* non-attendant
* severe anemia/micro nutrient deficiency
* thyroid disease
* medication/supplementation
* not willing to participate

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-07-28 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
To access the improvement in child Iron deficiency anemia | Will be accessed at Base-line (at start), Mid-line (after 4 months) and End-line (8 months)
  change in serum Hemoglobin, serum ferritin and serum transferrin receptors
To access the improvement in children Vitamin A status | Will be accessed at Base-line (at start), Mid-line (after 4 months) and End-line (8 months)
  Change in Serum retinol binding protein
To access the improvement in children Zinc status | Will be accessed at Base-line (at start), Mid-line (after 4 months) and End-line (8 months)
  Change in serum zinc

SECONDARY OUTCOMES:
Difference in the children anthropocentric status | Base-line (at start, 0 month), Mid-line (after 4 months) and End-line (8 months at start)
  Mean z-scores (weight-for-age, length-for-age z-scores, weight-for-length) based on the WHO child growth standards 2006
Effect on the household food security | Base-line (at start, 0 month), Mid-line (after 4 months) and End-line (8 months at start)
  Diet diversity score based on dietary intake and preferences by 24 hrs dietary recall and Household Food Security Scale
Enhancement in the early childhood development indicators | Base-line (at start, 0 month), Mid-line (after 4 months) and End-line (8 months at start)
  Gain change in the cognitive, motor and socio-emotional assessment through questionnaire filled by caretaker

CONTACTS AND LOCATIONS:
Overall Officials: Fakhar Gulzar, Principal Investigator — University of Veterinary and Animal Sciences, Lahore
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes